CLINICAL TRIAL: NCT07113873
Title: Clinical Performance of Ultra-translucent Multi-layer Monolithic Zirconia and Lithium Disilicate Ceramic Laminate Veneers
Brief Title: Patient Satisfaction and Clinical Performance of Ultra-translucent Multi-layer Monolithic Zirconia and Lithium Disilicate Ceramic Laminate Veneers. Randomized Control Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, MOHAMED ALI, dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Ultra Translucent Zirconia
Keywords: veneer; monolithic zirconia; lithium disilicate

STUDY DESIGN:
Intervention Model Description: zirconia monolithic ultra-translucent veneers
Who Masked: Participant
Masking Description: closed envelop
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lithium disilicate veneer (Active Comparator): After tooth preparation to receive conservative Emax veneers all preparation will be finished to provide smooth topography and allow maximum stability to the final restoration tooth surface and restoration surface will be treated according to the recommended protocol to attain best results
  Interventions: Other: lithium disilcate ceramics
- ultra translucent monolithic multi layered zirconia veneer (Experimental): Tooth preparation will be done using a turbine hand piece, minimal preparation will be resorted to by adopting the butt joint pattern that guarantees shortening the cutting edge to obtain the required translucent and esthetic aspect. The incisal edge will be prepared by depth guide stone; this will be followed by preparing the cervical region 0.1-0.3mm and the mid-region 0.3-0.5 mm The cutting edge will be reduced by 1.0-1.5 mm. After removing the enamel via a cone round-end stone to reach the required depth, the finishing lines will be adopting the light chamfer scheme. Moreover, the preparation will be extended to a labial surface without exceeding the interproximal contact, rounding all the edges and linear angles. Later,10 manufacturing the veneers will follow the exact laboratory steps for both the zirconia group.
  Interventions: Other: ultra-translucent monolithic multi layered zirconia

INTERVENTIONS:
Other: ultra-translucent monolithic multi layered zirconia — laminate veneer
  Arms: ultra translucent monolithic multi layered zirconia veneer
Other: lithium disilcate ceramics — laminate veneer
  Arms: lithium disilicate veneer

SUMMARY:
Despite of the improved esthetics of ultra-translucent zirconia, bonding between resin cement and zirconia is difficult to achieve because of their chemical inertness and lack of silica content. However, the effect of the bond strength with the new generation of high-translucent zirconia materials is not clear and further studies are needed. Kongkiatkamon, Suchada et al., (2023) The long-term bond strength of cubic zirconia was similar to 3Y-TZP zirconia and lithium disilicate ceramics and showed sufficient bond strength. A 5-mol% yttria-stabilized tetragonal Zr polycrystal showed high shear bond strength similar to Li disilicate glass-ceramic. Air blasting of Zr followed by primers and resin cements based on 10-MDP monomer has proven its efficiency in Zr-resin bonding. Both ultra-translucent 5Y-PSZ Zr and Li disilicate offer viable options for esthetic restorations on anterior teeth Adak et al. (2023),Elsisi et al. (2024) Currently, there is a lack of reports in the literature regarding the long-term clinical performance of ultra-translucent zirconia, especially considering its use in manufacturing monolithic veneers. Therefore, the purpose of the present clinical trial is to assess the validity of using ultra-translucent multi-layer zirconia ceramic veneer as an alternative to lithium disilicate ceramic veneer

DETAILED DESCRIPTION:
Preservation of tooth structure and prevention of needless tooth structure removal are basic and important principles in prosthodontics. Striving to achieve the cosmetic aspect is also a basic requirement, especially in the modern world Fawakhiri et al. (2023) Porcelain laminate veneers are one of the most popular cosmetic and minimally invasive dental treatments. These veneers can change the color, contour, shape, and size of the teeth they cover and bond to tooth structure with the use of adhesive cements. A thin layer of enamel (0.5-.8 mm) is removed to provide space for each veneer Piemjai and Donpinprai (2023) Several ceramic materials are currently indicated for veneers: lithium disilicate, feldspathic ceramic, feldspathic reinforced with leucite, fluorapatite, and lithium silicate reinforced with zirconia. All of these ceramics exhibit high translucency characteristics due to the high content of glassy matrix in their composition, thus providing highly satisfactory esthetics in addition to excellent adhesion to resin cement through the conditioning with hydrofluoric acid (4%-10%) followed by silanization Souza et al. (2017) Lithium disilicate ceramics belong to the silica-based ceramics family. They are commonly used for the fabrication of laminate veneers owing to their excellent optical properties, including their superior translucency and strong bonding to the tooth enamel surface when etched with hydrofluoric acid and then silanized Ojeda et al. (2023) Longevity is one of the most important factors to predict the survival and success of restorations. Many longitudinal clinical studies have evaluated the performance of ceramic veneer restorations and have confirmed good clinical performance, excellent aesthetics, and a high level of patient satisfaction. Major clinical complications commonly resulting in the failure of ceramic veneer restorations are fracture and debonding (Monaraks, 2018) The long-term clinical success of ceramic-based restorations is strongly dependent on their retention to teeth or abutment substrates by using adhesive systems and resin-matrix cements in vitro research has shown that load-to-fracture values of monolithic zirconia are higher than those of LS2; the latter, in turn, are higher than those of ZLS Zarone et al. (2019) ,(Souza et al., 2023) 6 The excellent biocompatibility and superior mechanical properties of zirconium dioxide (zirconia) ceramics make them a material of choice in prosthetic dentistry. Nevertheless, zirconia ceramics have not been used for the fabrication of laminate veneers because the opaqueness and low translucency of zirconia ceramics yield undesirable esthetic results. Due to the absence of any glassy matrix, zirconia is free from silica and, consequently, cannot be conditioned with conventional acid etching techniques, differently from glass-ceramics. Kusaba, Kosuke et al., (2018) , Zarone et al. (2019) Lately, the ultra-translucent multilayered zirconia has been introduced to the market. This material structured to replicate the naturality of teeth according to each anatomical region, keeping translucency at the incisal edge and a higher opacity at the cervical area. The multilayer blanks are pre-layered and thus contain different shades. There is scientific evidence reporting that the darker the color the higher the degree of opacity, that's to say the lower the translucency becomes. The color of the blanks is increasingly lighter and thus more translucent towards the incisal area. The dental technician can use CAD software to help to determine color sequences and intensities by positioning the constructed restoration in the blank. One advantage resulting from the combination of highly esthetic (color and translucency values are similar to those of natural teeth) and highly stable materials is better treatment with restorations with low space requirements. This Ultra-translucent Zirconia ceramic veneers have a minimum thickness of 0.1-0.3 mm, a more conservative option than glass-ceramic restorations Alqutaibi et al. (2022), Gomes et al., (2022), ("Three Generations of Zirconia: From Veneered to Monolithic. Part I.," 2017)

ELIGIBILITY:
Inclusion Criteria:

1- Age between 18 and 50 years. 2. Absence of abnormal functional habits such as bruxism. 3. Good condition of gingival and periodontal tissues. 4. Good oral health. 5. A clear indication for patients for treatment with ceramic laminate veneers: Presence of diastema, moderate discolored dental restorations, slight modification of color in the discolored teeth, and modification of shape and sizes of the teeth.

6. Patient commitment for attending follow up session

Exclusion Criteria:

1. Age under 18 years
2. Bad oral hygiene
3. Dysfunctional habits and bruxism
4. Periodontal diseases
5. High risk of caries
6. Inadequate enamel for bonding
7. Extreme staining and color change in tooth -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-01-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 24 month
  Numerical (discrete) ("0" unsatisfied - "10" satisfied)

SECONDARY OUTCOMES:
Color Stability | 24 month
  ΔE<2.7
Marginal Integrity | 24 month
  Alpha (A) No visible evidences of crevice along the margins; no catch or penetration of the explorer.
  * Bravo (B) Visible evidence of crevice and/or catch of explorer; no penetration of the explorer.
  * Charlie (C) Visible evidence of crevice and penetration of the explorer
Gingival Health | 24 month
  * Alpha (A) Normal gingiva
  * Bravo (B) Mild inflammation - slight change in color and slight edema but no bleeding on probing 11 13-Participant timeline
  The patient will be treated in a regular sequence:
  visit 1: proper examination for the participants (clinically and radiographically) and alginate impressions for diagnosis on primary casts and for mounting Visit 2: Preparation for abutment teeth, final impression using elastic impression material and provisional restoration.
  Visit 3: permanent cementation of the final restoration Visit 4: follow-up every 3month for 24 months 14-Calculated sample size: Sample size calculated depending on a previous study by Verniani et al. (2024) as reference. According to this study, the minimally accepted sample size was 7 per group, when mean ± standard deviation of patient satisfaction at baseline in-group I was 7.1±1.5 while after 2 years was 9.5 ±2, with 1.33 effect size, when the power was 80 % & type I error probability was 0.05. Total sample si
Retention | 24 month
  * Alpha (A)No loss of restorative material
  * Bravo (B) Partial loss of restorative material
  * Charlie (C) Missing restoration

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No